CLINICAL TRIAL: NCT03519139
Title: Individual Nutritional Intervention for the Prevention of Readmission Among Geriatric Patients - a Randomized Clinical Study
Brief Title: Individual Nutritional Intervention for the Prevention of Readmission Among Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-17039329
Record Dates: First submitted 2018-04-09; First posted 2018-05-08 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Readmission
Keywords: Geriatric patients, nutritional counselling, homevisit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individual dietary counselling (Experimental): three individual dietary counsellings. The first at the hospital by discharge, then in week 1 and week 3 at the subject's home/the respite care after discharge and, if necessary, telephone follow-up in weeks 2 and 4 after discharge
  Interventions: Other: individual dietary counselling
- Control (No Intervention): standard counselling provided by the hospital at discharge. The standard counselling may include nutritional prescription and nutritional plan, but no follow-up to the nutrition plan after the discharge.

INTERVENTIONS:
Other: individual dietary counselling — individual dietary counsellings with the aim to ensure sufficient coverage of energy and protein needs of the test subjects
  Arms: individual dietary counselling

SUMMARY:
The purpose of this study is to investigate whether a four-week individual nutritional intervention can reduce the readmission/hospitalization rate among geriatric patients who are discharged to their private home or respite care. Secondarily, whether an individual nutritional intervention can improve nutritional status, functional status, quality of life, muscle strength and reduce mortality in geriatric patients after discharge Two sub-points are investigated using feasibility studies - if photography documentation of meals can be used in practice to assess the energy and protein intake of geriatric patients and whether photography documentation of the refrigerator content at first home visits in the intervention group can predict whether there is an increased risk of readmission.

DETAILED DESCRIPTION:
Method/Design:

The trial is conducted as a randomized clinical trial, with recruitment of 40 medical geriatric patients (definition: ≥65 years of age with at least two diagnoses, e.g. hypertension, cardiovascular diseases, diabetes, chronic obstructive pulmonary disease, rheumatic diseases or apoplexy). At discharge the test subjects are randomized to receive either individual dietary counseling or standard treatment with follow-up 30 and 60 days after discharge. All data are collected prior to randomization. The intervention consists of three individual dietary counsellings with the aim to ensure sufficient coverage of energy and protein needs of the subjects (the first at the hospital by discharge, then in week 1 and week 3 at the subject's home/the respite care after discharge) and, if necessary, telephone follow-up in weeks 2 and 4 after discharge. The intervention group, if possible, are asked to take photos of all they eat and drink for two days before individual dietary counselling and send the photos electronically to the responsible investigators before the meeting.

Recruitment:

Only admitted patients are included in the trial. Attending physician finds the patients through the Health Platform at Sydsjællands University Hospital. The care staff or the attending physician asks whether the patient is willing to talk with the responsible investigators. The responsible investigators then make personal contact with the geriatric patients while they are hospitalized. Patients will be informed orally and in writing about the trial of the responsible investigators. Patients also receive pamphlets about test subjects rights in a health science research project published by the National Science Ethics Committee with the purpose of giving patients an informed basis to make a decision.

Patients are informed that they can take a family member or friend to the next conversation. Patients receive at least 24 hours of deliberation time, after which they are contacted by the responsible investigators. Patients who wish to participate in the trial are asked to sign a consent statement. This statement is also signed by the responsible investigator who has given the patient oral information about the trial. The subjects are offered a copy of the consent statement. To ensure uninterrupted conversation, conversation will take place in a room without other people or alternatively in the patient's room and a partition will be put of if the patient is not in a room by them self.

Patients who meet the inclusion criteria, wishes to participate in the trial and have signed the consent statement will be contacted again on the date of discharge or the day before, where the trial starts. Test subject may at any time, orally, in writing or by other clear indication, withdraw their consent for participation and withdraw from the trial.

Sample size:

Based on the primary output "readmission/hospitalization of geriatric patients within a month", the sample size is estimated to be at least 20 subjects in the intervention and control groups, respectively. A total of at least 40 subjects.

Statistical analysis:

Hypothesis testing will take place using nonparametric statistical tests, as the data can not be assumed to be normal distribution (Mann-Whitney U and Wilcoxon). Fisher's exact test [M1] is used for analysis of categorical data. Correlations are analyzed using Spermann analysis

ELIGIBILITY:
Inclusion Criteria:

* recruited at Medical Department at Sjælland University Hospital, Køge (sections M1, M2, M6, L1) and discharged to one of following municipalities: Greve, Køge, Roskilde, Solrød and Stevns
* geriatric patients according to the definition
* competent adult and Danish speaking who are able to give written consent
* oral nutrition possible (no tube feeding or intravenous nutrition)
* discharged planned for home or respite care or similar (e.g. family).

Exclusion Criteria:

* diagnosed dementia or under investigation for dementia
* nursing home resident or discharged to nursing homes
* terminal patients
* patients who desire weight loss
* scheduled readmission.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
readmission-or hospitalization rate (%) | 30 days after discharge
  readmission for the same diagnosis as at discharge. Hospitalization for a new diagnosis

SECONDARY OUTCOMES:
readmission-/hospitalization rate (%) | 60 days after discharge
  readmission for the same diagnosis as at discharge. Hospitalization for a new diagnosis
number of days between readmission or hospitalization and discharge (days) | 30 and 60 days after discharge
  date minus date
nutritional status (%) | 30 and 60 days after discharge
  The proportion of subject who has covered at least 75% of estimated energy and protein needs
functional status (score, points) | 30 and 60 days after discharge
  Functional recovery score: P-ADL, I-ADL and mobility
Quality of Life (score, points) | 30 and 60 days after discharge
  EQ-5D-5L
muscle strenght (dyn) | 30 and 60 days after discharge
  Hand-grip strenght

OTHER OUTCOMES:
mortality (%) | 30 and 60 days after discharge
  % died from any cause
side effects in connection with the intervention (number) | 30 and 60 days after discharge
  any side-effects reported

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, ass. prof., Principal Investigator — University of Copenhagen
Locations (1):
- Sjaellands Universitetshospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Yes
anonymised individual participant data for primary and secondarily outcomes measurement will be made available
Supporting Information: Study Protocol
Time Frame: data will be available within one year of study completion
Access Criteria: Author or co-author from the University of Copenhagen

REFERENCES:
- [Derived] Cramon MO, Raben I, Beck AM, Andersen JR. Individual nutritional intervention for prevention of readmission among geriatric patients-a randomized controlled pilot trial. Pilot Feasibility Stud. 2021 Nov 15;7(1):206. doi: 10.1186/s40814-021-00926-9. PMID 34782015